CLINICAL TRIAL: NCT02153450
Title: A Pilot Trial of Stereotactic Body Radiation Therapy and Metformin for Borderline-Resectable and Locally-Advanced Pancreatic Adenocarcinomas
Brief Title: Stereotactic Radiosurgery and Metformin in Patients With Borderline-Resectable or Locally-Advanced Pancreatic Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4213; NCI-2014-01172 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 4213 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage I-III Pancreatic Cancer
Keywords: pancreatic cancer; Radiation; Metformin; Pancreatic Adenocarcinomas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Metformin; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (stereotactic radiosurgery, metformin hydrochloride) (Experimental): Patients receive metformin hydrochloride PO daily or BID on days -11 to -1. Patients then undergo stereotactic radiosurgery 5 days a week for 5 weeks and receive concurrent metformin hydrochloride* PO BID for 5 weeks. Patients undergo laparotomy on week 6 (or weeks 5-7). Systemic therapy continues as soon as it is considered feasible by the treating physicians.
  *NOTE: Metformin hydrochloride should be stopped 2 days before laparotomy.
  Interventions: Drug: metformin hydrochloride; Radiation: stereotactic radiosurgery

INTERVENTIONS:
Drug: metformin hydrochloride — Given PO
  Other Names: Glucophage
Radiation: stereotactic radiosurgery — Undergo stereotactic radiosurgery

SUMMARY:
This pilot clinical trial studies stereotactic radiosurgery and metformin hydrochloride in treating patients with pancreatic cancer that may be removed (borderline-resectable) or not removed by surgery. Stereotactic radiosurgery may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Metformin hydrochloride, used for diabetes, may also kill cancer cells as demonstrated in laboratory studies. Giving stereotactic radiosurgery with metformin hydrochloride may kill more tumor cells.

DETAILED DESCRIPTION:
This is an open label pilot, single-center, non-randomized trial is designed to evaluate the tolerability and preliminary activity of the combination of stereotactic body radiation therapy (SBRT) with metformin for resectable and locally-advanced pancreatic/periampullary cancers.

PRIMARY OBJECTIVES:

The primary objectives of this study are to:

1) To determine if the addition of metformin to SBRT adds minimal additional toxicity for patients with A). borderline-resectable or B). not surgically resectable pancreatic adenocarcinomas.

SECONDARY OBJECTIVES:

I. Evaluate the clinical/pathological response and resectability rates associated with these regimens.

OUTLINE:

Patients receive metformin hydrochloride orally (PO) daily or twice daily (BID) on days -11 to -1. Patients then undergo stereotactic radiosurgery 5 days a week for 5 weeks and receive concurrent metformin hydrochloride* by mouth, two times a day for 5 weeks. Patients undergo laparotomy on week 6 (or weeks 5-7). ). Systemic therapy continues as soon as it is considered feasible by the treating physicians.

*NOTE: Metformin hydrochloride should be stopped 2 days before laparotomy.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to provide written informed consent
* Histologically and/or cytologically confirmed adenocarcinoma of the pancreas, clinical stage T1-4, N0-1, M0
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Hemoglobin ≥ 9.0 g/dl
* Alkaline phosphatase < 3 x upper limit of normal (ULN)
* Albumin > 2.5 g/dL
* Absolute neutrophil count ≥ 1500/mm^3
* Platelet count ≥ 75,000/mm^3
* Total bilirubin < 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) ≤ 2.5 x institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 x institutional upper limit of normal
* Creatinine ≤ 1.5
* Borderline-resectable or locally-advanced pancreatic cancer (based upon impression of the surgical oncologist, in conjunction with radiologic consultations) as defined per the Alliance consensus :

  * Borderline-resectable

    * An interface between the primary tumor and superior mesenteric vein (SMV)/portal vein measuring 180 degrees or greater of the circumference of the vein wall
    * Short-segment occlusion of the SMV/portal vein but with suitable vessel proximal and distal to the obstruction to allow safe resection and reconstruction
    * Short-segment interface (of any degree) between the tumor and the hepatic artery with normal artery proximal and distal to the interface that is amenable to resection and arterial reconstruction
    * An interface between the tumor and the SMA or celiac trunk measuring less than 180 degrees of the circumference of the artery wall
  * Not surgically resectable due to one or more of the following things

    * Patient is not a surgical candidate due to medical comorbidities and/or poor performance status
    * Patient elects not to undergo surgical therapy
    * Patient has locally-advanced pancreatic cancer based on having one of the following:

      * Encasement of the SMA/celiac artery (>180 degrees).
      * Involvement of the SMV/portal vein without options for reconstruction.
      * Aortic invasion or encasement.
* Women of child-bearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) 6 weeks prior to study entry, for the duration of study participation and for 6 months after completing treatment; should a woman become pregnant or suspect that she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately
* Patients previously treated with chemotherapy are eligible unless they have evidence of local or distant disease progression; patients must have completed their last cycle of chemotherapy at least two weeks prior to study enrollment
* Patients currently taking metformin are eligible for participation.
* Women of child-bearing potential and male patients who are sexually-active must agree to use effective methods of birth control throughout protocol treatment.
* Patients must not have poorly-controlled diarrhea (no more than 4 loose stools per day). Patients may be reconsidered for the study if the diarrhea resolves.

Exclusion Criteria:

* Evidence of gross duodenal invasion, gastric outlet obstruction
* Gastrointestinal perforation or intra-abdominal abscess (< 3 months); recent (< 3 months) gastrointestinal (GI) bleeding from gastric or duodenal ulcer
* Systemic collagen vascular disease including scleroderma or systemic lupus erythematosus (SLE); rheumatoid arthritis is eligible
* Serious active infection requiring intravenous (IV) antibiotics
* Conditions leading to inadequate gastrointestinal tract absorption as determined by the treating physician and/or investigator
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Poorly-controlled diarrhea (> 4 loose bowel movement [BM]/day without use of anti-motility agents) within 7 days of study enrollment; patients may be reconsidered for the study if the diarrhea resolves
* Comorbid conditions that, in the opinion of the investigator, would complicate safety or compliance such as known human immunodeficiency virus (HIV) or current substance abuse
* Patients who are pregnant or lactating
* Patients who are unwilling or unable to comply with study and/or follow-up procedures
* Treatment for other carcinomas within the last two years, except cured non-melanoma skin cancer, curatively treated in-situ cervical cancer, or localized prostate cancer with stable prostate-specific antigen (PSA)
* Multi-focal pancreatic lesions concerning for cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2020-06-13 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) rate scored according to the National Cancer Institute Common Toxicity Criteria version 4 | Up to 21 days post-treatment
  The rate of DLT for each treatment group will be estimated based on the number of incidences using a binomial distribution and its confidence intervals will be estimated using Wilson's method. The factors associated with DLT will be identified using logistic regression using forward model selection procedure

SECONDARY OUTCOMES:
Clinical response rate using the revised Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 2 years
  Using a binomial distribution and its confidence intervals will be estimated using Wilson's method.
Progression-free survival using the revised RECIST version 1.1 | Time from start of treatment to time of progression or death, whichever occurs first, assessed up to 2 years
  The factors associated with progression-free survival will be identified using logistic regression using forward model selection procedure.
Overall survival | Up to 2 years
  The probability of overall survival along with median survival for each treatment group will be estimated using Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Dorth, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States